CLINICAL TRIAL: NCT01260532
Title: The Association of Costimulatory Molecules and PPAR-polymorphisms With Autoimmune Thyroid Disease in Taiwan
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Jiunn-Diann Lin, Division of Endocrinology and Metabolism
Other Study IDs: 98049
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2010-12-15 (Estimated); Status verified 2010-12

CONDITIONS: AITd Patients With Different Polymorphisms
Keywords: Autoimmune thyroid disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Graves' disease: no intervention
- Hashimoto's thyroiditis: no intervention
- Healthy subjects: no intervention

SUMMARY:
Autoimmune thyroid disease is the most common organ-specific autoimmune disease. AITD include Graves' disease and Hashimoto's thyroiditis. Although the pathogenesis of AITD remains unclear, it is generally thought that the mechanisms of the disease is a complex disease in which susceptibility genes and environmental triggers act in concert to initiate the autoimmune response to the thyroid.

The initial step of thyroid autoimmunity is the activation of T cells. The activation of T cell requires two signals: firstly, thyroid follicular cells or antigen presenting cells binds to T cell receptor through antigenic HLA complex. Secondly, the activation of T cells is also required the interaction of costimulatory molecules between thyroid follicular cells and immune cells, including CTLA-4, CD 40, CD28, ICOS. PPAR- is a kind of intranuclear transcription factor, associated with adipogenesis and inflammation. Some reports showed that PPAR- polymorphism may have a protective effect from Graves' ophthalmopathy.

The goal of the study is to investigate the relationship among SNP and mRNA of costimulatory molecules and PPAR- , serum cytokine including TNF- and sIL-2R, and clinical characteristics in AITD patients. From the study, we hope to clarify the role of costimulatory molecules and PPAR- polymorphism in AITD.

DETAILED DESCRIPTION:
Autoimmune thyroid disease is the most common organ-specific autoimmune disease. AITD include Graves' disease and Hashimoto's thyroiditis. Although the pathogenesis of AITD remains unclear, it is generally thought that the mechanisms of the disease is a complex disease in which susceptibility genes and environmental triggers act in concert to initiate the autoimmune response to the thyroid.

The initial step of thyroid autoimmunity is the activation of T cells. The activation of T cell requires two signals: firstly, thyroid follicular cells or antigen presenting cells binds to T cell receptor through antigenic HLA complex. Secondly, the activation of T cells is also required the interaction of costimulatory molecules between thyroid follicular cells and immune cells, including CTLA-4, CD 40, CD28, ICOS. PPAR- is a kind of intranuclear transcription factor, associated with adipogenesis and inflammation. Some reports showed that PPAR- polymorphism may have a protective effect from Graves' ophthalmopathy.

The goal of the study is to investigate the relationship among SNP and mRNA of costimulatory molecules and PPAR- , serum cytokine including TNF- and sIL-2R, and clinical characteristics in AITD patients. From the study, we hope to clarify the role of costimulatory molecules and PPAR- polymorphism in AITD.

ELIGIBILITY:
Inclusion Criteria:

* Autoimmune thyroid patients
* patients who cut Nodular Goiter in Wanfang Hospital

Exclusion Criteria:

* none

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Autoimmune thyroid patients
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-07; Study Completion 2019-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jiunn-Diann Lin, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan